CLINICAL TRIAL: NCT00324025
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Mycograb® as Adjunctive Therapy for Cryptococcal Meningitis in Patients With AIDS
Brief Title: Efficacy and Safety of Mycograb as Adjunctive Therapy for Cryptococcal Meningitis in Patients With AIDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MYC123A2202; NTP/Mycograb/003A; NCT00804635 (obsolete NCT alias)
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Cryptococcal Meningitis
Keywords: Cryptococcal meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — efungumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental): Mycograb
  Interventions: Drug: Mycograb
- 2 (Active Comparator): biological
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mycograb
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, multicenter efficacy and safety trial to evaluate Mycograb®. Subjects will be randomized to receive either Mycograb® (dosed 1 mg/kg) or placebo during the first week of induction therapy (amphotericin B plus 5-flucytosine) via a central line or peripheral venous line twice daily for 7 consecutive days. The total duration of the study will be approximately 24 months.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, parallel-group clinical trial is designed to evaluate Mycograb® versus placebo as adjunctive therapy to antifungal induction therapy (amphotericin B plus 5-flucytosine) in subjects who have acute cryptococcal meningitis associated with AIDS. After pre-study screening and baseline assessments and meeting all inclusion criteria, on Day 1 subjects will be randomized to 1 of 2 treatment arms:

Amphotericin B (conventional at 0.7 mg/kg, i.v. once daily) plus 5-flucytosine (100 mg/kg orally daily, divided QID), with placebo.

Amphotericin B (conventional at 0.7 mg/kg, i.v. once daily) plus 5-flucytosine (100 mg/kg orally daily, divided QID), with Mycograb®.

Study medication will be administered via a central line or peripheral venous line twice daily for 7 consecutive days (Days 1-7). A lumbar puncture with CSF culture colony counts, India ink microscopy, and measurement of cryptococcal antigen (CrAg) will be performed at Baseline, Days 3, 7, and 14,. CSF will also be assayed for concentrations of Mycograb® on Days 3, 7, and 14. The primary efficacy parameter will be the proportion of subjects considered cured at day 14 (combined clinical AND mycological outcome).

A complimentary clinical trial will be run in parallel with this study in South America and South Africa. The protocol used will be essentially as described here except that there will be an additional (3rd) treatment arm (Amphotericin B [conventional at 0.7 mg/kg, i.v. once daily}with Mycograb®)..

An interim analysis will be performed after 30 patients (US and/or non-US) have completed Day 14, for the following reasons:

To evaluate the safety of Mycograb® by reviewing the adverse events classified by the investigator as possibly related to the study drug To adjust the proposed sample size if necessary. A Safety Monitoring Committee and an independent expert will assess the safety profile of Mycograb®.

A total of 40 completed patients are planned for the US. It is estimated that enrollment will require 54 screened and 48 enrolled to achieve 40 completed patients. The total duration of the trial will be approximately 24 months. If the recruitment rate is low in the US, the number from the US may be reduced, having been replaced by patients outside the US where cryptococcosis is more prevalent.

ELIGIBILITY:
Inclusion criteria:

Male or non-pregnant female who is >18 years old, HIV-positive or unknown, with acute, either first or recurrent episode of cryptococcal meningitis Currently on no treatment, or receiving treatment (< 3 days) with either amphotericin B plus 5-flucytosine, or amphotericin B alone. Positive CSF culture for Cryptococcus neoforman. Physical signs and symptoms of meningitis, evidenced by one or more of the following: fever, headache, meningeal signs and neurologic findings.

Exclusion criteria:

Excluded for coma, or significant other medical conditions. Subject has other opportunistic fungal infections that requires other systemic antifungal therapies.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
proportion of patients cured (combined clinical and microbiological response) versus placebo | Day 14

SECONDARY OUTCOMES:
Safety of Mycograb versus placebo. Safety assessment will include: physical examination, vital signs, laboratory parameters, adverse events, serious adverse events. | Week 10
Assess the cerebrospinal fluid (CSF) penetration of Mycograb | Days 3, 7 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, MD, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - University of Alabama School of Medicine, Birmingham, Alabama
  - Department of Medicine/Infectious Disease, MC 7881, University of Texas Health Science Center, San Antonio, Texas